CLINICAL TRIAL: NCT06953583
Title: A Phase 3, 2-Part, Randomized, Double-Blind, Placebo-Controlled Study (Part 1) and Open-Label Extension (Part 2) to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Omaveloxolone (BIIB141) in Participants With Friedreich's Ataxia Aged 2 to < 16 Years
Brief Title: A Study to Learn More About the Effects and Long-Term Safety of BIIB141 (Omaveloxolone) in Participants With Friedreich's Ataxia Aged 2 to 15 Years Old (BRAVE)
Acronym: BRAVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 296FA301; 2025-520896-13 (Other: EU CT Number)
Record Dates: First submitted 2025-04-11; First posted 2025-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — omaveloxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 of the study is placebo-controlled and Part 2 is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 RCT: Omaveloxolone (Experimental): Participants will receive a single oral dose of omaveloxolone once a day (QD) for up to 52 weeks in Part 1 of the study.
  Interventions: Drug: Omaveloxolone
- Part 1 RCT: Placebo (Placebo Comparator): Participants will receive placebo, orally, QD for up to 52 weeks in Part 1 of the study.
  Interventions: Drug: Placebo
- Part 2 OLE: Omaveloxolone (Experimental): Participants who complete Part 1 of the study and are eligible will receive a single oral dose of omaveloxolone, QD for up to 104 weeks in the Part 2 OLE study.
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm.
  Other Names: BIIB141, SKYCLARYS, RTA-408
  Arms: Part 1 RCT: Omaveloxolone; Part 2 OLE: Omaveloxolone
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part 1 RCT: Placebo

SUMMARY:
In this study, researchers will learn more about the effects and safety of BIIB141, also known as omaveloxolone or SKYCLARYS®. This drug has been approved, or made available for doctors to prescribe, for people with Friedreich's Ataxia (FA) who are at least 16 years old. But, it is not yet available for children and teens with FA who are younger than 16 years old. The main objective of this study is to learn how BIIB141 works in the body and about its safety in children and teens who are 2 to 15 years old.

The main questions researchers want to answer in this study are:

* How does BIIB141 affect the participants' FA symptoms balance and stability?
* How many participants have medical problems during the study?
* Are there any changes in the participants' overall health during the study?
* Are there any changes in the participants' heart health?
* Are there any changes in how the participants move through puberty? Puberty is the time in someone's life when their body changes from a child to an adult.

Researchers will also learn more about:

- How the body processes BIIB141 in children and teens

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into their study research center.
* There are 2 parts in this study. During Part 1, participants will take either BIIB141 or a placebo once a day.
* In Part 1, participants will take BIIB141 or the placebo in a study research center on Day 1, and then at in-person visits at Week 4, Week 12, Week 26, and Week 52. On all other days, they will take BIIB141 or the placebo at home. Part 1 lasts up to 52 weeks.
* During Part 2, participants from Part 1 will either continue taking BIIB141 or start it if they were taking the placebo. Part 2 will last up to 104 weeks.
* In Part 1, participants will have up to 10 visits to their study research center and a phone call at Week 2. In Part 2, participants will have visits at Weeks 4, 8,12, 26, and every 26 weeks after that until they leave the study, and a phone call at Week 2. There will be a final phone call to check on the participants' health 31 days after their last dose.
* Each participant will be in the study for up to about 3 years

DETAILED DESCRIPTION:
The primary objective of Part 1 randomized controlled trial (RCT) is to evaluate the efficacy of omaveloxolone at Week 52 and the secondary objectives are to evaluate safety of omaveloxolone through Week 52 and the concentration of omaveloxolone after single and multiple dose administration. The primary objective of Part 2 open-label extension (OLE) trial is to evaluate the safety and tolerability of long-term omaveloxolone use and the secondary objective is to evaluate the efficacy of omaveloxolone following long-term use.

ELIGIBILITY:
Part 1 RCT: Key inclusion criteria:

* Diagnosed with genetically confirmed Friedreich's Ataxia (FA), i.e., homozygous for guanine-adenine-adenine (GAA) repeat expansion in intron-1 of the frataxin gene, or GAA repeat expansion in 1 allele and with point mutations or deletions, or other non-GAA expansion mutations in the other allele.
* Symptomatic for FA as confirmed by clinician assessment. a. Children 7 to < 16 years must also have an upright stability score (USS) score of 10 to ≤ 34 at baseline

Part 1 RCT: Key exclusion criteria:

* Glycosylated hemoglobin A1C (HbA1c) > 11%
* B-type natriuretic peptide (BNP) > 200 picograms per milliliter (pg/mL) at screening
* Ejection fraction (EF) < 40% [based on echocardiogram (ECHO) performed at screening visit]
* Clinically significant cardiac disease except mild to moderate cardiomyopathy

Part 2 OLE: Eligibility criteria:

* Participants have completed Part 1 RCT of the study and no discontinuation criteria have been met
* Safety and tolerability data from Part 1 RCT are supportive of continuation in the judgement of the investigator

  1. If BNP is > 200 pg/mL at the previous visit assessment, Part 2 Day 1 should be delayed until BNP is < 200 pg/mL.
  2. If any other clinically significant laboratory abnormalities are present based on the previous visit assessments, Part 2 Day 1 should be delayed until the abnormalities are resolved.
  3. In the event of intercurrent illness or other change in health status of the participant, additional Part 1 screening assessments may be repeated prior to initiation of Part 2, based on the judgement of the investigator in consultation with the medical monitor.
  4. If dosing has been interrupted at the end of Part 1, Part 2 Day 1 should be delayed until resumption of study drug treatment is appropriate per Section 8.2.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-11-16 (Estimated); Study Completion 2029-11-22 (Estimated)

PRIMARY OUTCOMES:
Part 1 RCT: Change From Baseline in Upright Stability Score (USS) Subscale E of Modified Friedreich's Ataxia Rating Scale (mFARS) | Baseline, Week 52
  The mFARS is a validated and sensitive rating scale that was developed to quantitatively assess the severity of the neurologic features of FA in adults and adolescents. Scores on the mFARS range from 0 to 93, with lower scores indicating better neurological function. The subscales of the mFARS assessment and maximum score for each subscale are: bulbar function (Subscale A; 2 assessments of speech and cough; maximum score = 5), upper limb coordination (Subscale B; 5 assessments of coordination of movement and function in arms and hands with each limb scored individually; maximum score = 36), lower limb coordination (Subscale C; 2 assessments of coordination of movement and function of lower limbs with each limb scored individually; maximum score = 16), and upright stability (USS, Subscale E; 9 assessments of sitting posture, stance, tandem walk, and gait assessments; maximum score = 36).
Part 2 OLE: Number of Participants With Treatment-Emergent Adverse Event (TEAE) and Treatment-Emergent Serious Adverse Event (TESAE) | From the first dose of the study drug in Part 2 up to the end of follow-up period in Part 2 (up to Week 105)
Part 2 OLE: Number of Participants With Change From Baseline in Cardiac Function Assessed by Echocardiogram (ECHO) | Baseline (Week 52) up to Week 104
Part 2 OLE: Change From Baseline in Height | Baseline (Week 52) up to Week 104
Part 2 OLE: Change From Baseline in Weight | Baseline (Week 52) up to Week 104
Part 2 OLE: Change From Baseline in Body Mass Index (BMI) | Baseline (Week 52) up to Week 104
Part 2 OLE: Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline (Week 52) up to Week 104
  The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed to assess severity and track suicidal events through any treatment of individuals ≥ 6 years of age. The C-SSRS is a clinical interview providing a summary of both ideation and behavior that can be administered by the clinician during any evaluation or risk assessment to identify the level and type of suicidality present. The assessment includes "yes" or "no" responses for 5 questions each, related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings are provided for severity of ideation, from 1 to 5, with 5 being the most severe.
Part 2 OLE: Percentage of Participants at Each Tanner Stage | Baseline (Week 52) up to Week 104
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected at baseline for all participants and will be stopped once the participant reaches Tanner Stage 5 in all gender-appropriate scales.
Part 2 OLE: Number of Participants at Each Tanner Stage | Baseline (Week 52) up to Week 104
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected at baseline for all participants and will be stopped once the participant reaches Tanner Stage 5 in all gender-appropriate scales.

SECONDARY OUTCOMES:
Part 1 RCT: Change From Baseline in Friedreich's Ataxia-Health Index (FA-HI) | Baseline, Week 52
  The FA-HI is a participant reported survey that assesses overall disease burden on a 100-point scale, with 0 representing no disease burden and 100 representing the maximum level of disease burden containing 113 symptoms questions representing 18 symptomatic subscales.
Part 1 RCT: Change From Baseline in Modified Friedreich's Ataxia Rating Scale (mFARS) | Baseline, Week 52
  The mFARS is a validated and sensitive rating scale that was developed to quantitatively assess the severity of the neurologic features of FA in adults and adolescents. Scores on the mFARS range from 0 to 93, with lower scores indicating better neurological function. The subscales of the mFARS assessment and maximum score for each subscale are: bulbar function (Subscale A; 2 assessments of speech and cough; maximum score = 5), upper limb coordination (Subscale B; 5 assessments of coordination of movement and function in arms and hands with each limb scored individually; maximum score = 36), lower limb coordination (Subscale C; 2 assessments of coordination of movement and function of lower limbs with each limb scored individually; maximum score = 16), and upright stability (USS, Subscale E; 9 assessments of sitting posture, stance, tandem walk, and gait assessments; maximum score = 36).
Part 1 RCT: Change From Baseline in Patient Global Impressions-Severity (PGI-S) | Baseline, Week 52
  PGI-S will be conducted for participants 7 to < 16 years of age. These are clinically meaningful outcome measures that are participant-relevant across all age groups and disease severities for this population. PGI -S is a 1-item questionnaire where the response is recorded on a 4-point scale scored as: 1-normal, 2-mild, 3-moderate, or 4-severe.
Part 1 RCT: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) | Baseline, Week 52
  The CGI-S will be conducted for all enrolled participants, 2 to < 16 years of age. The CGI-S rating evaluates the severity of individual symptoms and treatment response in participants with mental disorders. The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Part 1 RCT: Change From Baseline in Friedreich's Ataxia-Activities of Daily Living (FA-ADL) | Baseline, Week 52
  Participants will answer the 9 questions of the FA-ADL survey in an interview style conducted by any site staff. The FA-ADL survey assesses 9 concepts: (1) speech; (2) swallowing; (3) cutting food and handling utensils; (4) dressing; (5) personal hygiene; (6) falling; (7) walking; (8) quality of sitting position; and (9) bladder function.
Part 1 RCT: Number of Participants With Treatment-Emergent Adverse Event (TEAE) and Treatment-Emergent Serious Adverse Event (TESAE) | From first dose of study drug up to end of follow up period in Part 1 RCT (up to Week 54)
Part 1 RCT: Number of Participants With Change From Baseline in Cardiac Function Assessed by Echocardiogram (ECHO) | Baseline, Weeks 26 and 52
Part 1 RCT: Change From Baseline in Height | Baseline up to Week 52
Part 1 RCT: Change From Baseline in Weight | Baseline up to Week 52
Part 1 RCT: Change From Baseline in Body Mass Index (BMI) | Baseline up to Week 52
Part 1 RCT: Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline up to week 52
  The C-SSRS is a low-burden measure of the spectrum of suicidal ideation and behavior that was developed to assess severity and track suicidal events through any treatment of individuals ≥ 6 years of age. The C-SSRS is a clinical interview providing a summary of both ideation and behavior that can be administered by the clinician during any evaluation or risk assessment to identify the level and type of suicidality present. The assessment includes "yes" or "no" responses for 5 questions each, related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings are provided for severity of ideation, from 1 to 5, with 5 being the most severe.
Part 1 RCT: Percentage of Participants at Each Tanner Stage | Screening and Week 52
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected at baseline for all participants and will be stopped once the participant reaches Tanner Stage 5 in all gender-appropriate scales.
Part 1 RCT: Number of Participants at Each Tanner Stage | Screening and Week 52
  Assessment of Tanner stages (a scale of physical development) will be performed by a medical doctor experienced with this assessment. Tanner score ranges from Stage 1 (childhood) to Stage 5 (full physical maturity). Information regarding Tanner staging will be collected at baseline for all participants and will be stopped once the participant reaches Tanner Stage 5 in all gender-appropriate scales.
Part 1 RCT: Plasma Concentrations of Omaveloxolone | Pre-dose and post-dose on Day 1, Weeks 4, 12 and 26
Part 2 OLE: Change From Baseline in Modified Friedreich's Ataxia Rating Scale (mFARS), Including Upright Stability Score (USS) | Baseline (Week 52) up to Week 104
  The mFARS is a validated and sensitive rating scale that was developed to quantitatively assess the severity of the neurologic features of FA in adults and adolescents. Scores on the mFARS range from 0 to 93, with lower scores indicating better neurological function. The subscales of the mFARS assessment and maximum score for each subscale are: bulbar function (Subscale A; 2 assessments of speech and cough; maximum score = 5), upper limb coordination (Subscale B; 5 assessments of coordination of movement and function in arms and hands with each limb scored individually; maximum score = 36), lower limb coordination (Subscale C; 2 assessments of coordination of movement and function of lower limbs with each limb scored individually; maximum score = 16), and upright stability (USS, Subscale E; 9 assessments of sitting posture, stance, tandem walk, and gait assessments; maximum score = 36).
Part 2 OLE: Change From Baseline in Friedreich's Ataxia-Activities of Daily Living (FA-ADL) | Baseline (Week 52) up to Week 104
  Participants will answer the 9 questions of the FA-ADL survey in an interview style conducted by any site staff. The FA-ADL survey assesses 9 concepts: (1) speech; (2) swallowing; (3) cutting food and handling utensils; (4) dressing; (5) personal hygiene; (6) falling; (7) walking; (8) quality of sitting position; and (9) bladder function. Every participant will be instructed to answer the 9 questions. Total scores on FA-ADL will be used as a secondary endpoint to assess efficacy in participants 7 to < 16 years of age.
Part 2 OLE: Change From Baseline in Friedreich's Ataxia-Health Index (FA-HI) | Baseline (Week 52) up to Week 104
  The FA-HI is a participant reported survey that assesses overall disease burden on a 100-point scale, with 0 representing no disease burden and 100 representing the maximum level of disease burden containing 113 symptoms questions representing 18 symptomatic subscales.
Part 2 OLE: Change From Baseline in Patient Global Impressions-Severity (PGI-S) | Baseline (Week 52) up to Week 104
  PGI-S will be conducted for participants 7 to < 16 years of age. These are clinically meaningful outcome measures that are participant relevant across all age groups and disease severities for this population. PGI -S is a 1-item questionnaire where the response is recorded on a 4-point scale scored as: 1-normal, 2-mild, 3-moderate, or 4- severe.
Part 2 OLE: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) | Baseline (Week 52) up to Week 104
  The CGI-S will be conducted for all enrolled participants, 2 to < 16 years of age. The CGI-S rating evaluates the severity of individual symptoms and treatment response in participants with mental disorders. The CGI-S is a 7-point scale that that requires the clinician to rate the severity of the participant's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (34):
- United States (7):
  - UCLA Neurology Outpatient Clinic at Westwood, Los Angeles, California
  - Norman Fixel Institute for Neurological Diseases UF Health, Gainesville, Florida
  - USF Health Morsani College of Medicine Department of Neurology, Tampa, Florida
  - Children's Hospital of Philadelphia - Buerger Center for Advanced Pediatric Care - PIN, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital - PIN, Memphis, Tennessee
  - CHKD's Health Center - South Campus - PIN, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Murdoch Childrens Research Institute (MCRI), Parkville, Victoria
- Universitätsklinikum Innsbruck, Innsbruck, Austria
- Brazil (3):
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda - ME, Brasília, Federal District
  - University of Campinas (UNICAMP) School of Medical Sciences, Campinas, São Paulo
  - PSEG Centro de Pesquisa Clinica, São Paulo, São Paulo
- Canada (2):
  - McGill University, Montreal, Quebec
  - CHU de Quebec -Universite Laval, Québec, Quebec
- Rigshospitalet - Juliane Marie Centret (JMC) Copenhagen, Copenhagen, Denmark
- France (2):
  - CHU de Montpellier- Hôpital Gui De Chauliac, Montpellier, Hérault
  - AP-HP - Hôpital Armand Trousseau, Paris
- Germany (3):
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - UKGM - Universitätsklinikum Giessen und Marburg GmbH - Standort Gießen, Giessen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi, National Capital Territory of Delhi, India
- CHI at Temple Street, Dublin, Ireland
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome, Lazio
  - IRCCS Eugenio Medea - Polo. Scientifico Veneto, Conegliano, Veneto
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- King Faisal Specialist Hospital & Research Centre, Riyadh, Ar Riya, Saudi Arabia
- Spain (2):
  - Hospital Sant Joan de Deu - PIN, Espluges de Llobregat, Barcelona
  - Hospital Universitario La Paz - PPDS, Madrid
- Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Sheffield Children's Hospital - PPDS, Sheffield, South Yorkshire
  - University College London, Institue of Neurology, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org

REFERENCES:
- See also: Related Info — https://www.braveresearchstudy.com